CLINICAL TRIAL: NCT04500431
Title: Clinical Study to Evaluate the Safety and Feasibility of Targeting CD269 Chimeric Antigen Receptor Engineered T Cell (spCART-269) Injection in the Treatment of CD269-positive Multiple Myeloma
Brief Title: Clinical Study to Evaluate the Safety and Feasibility of spCART-269 Injection in the Treatment of MM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Aibin Liang，MD，Ph.D., Vice President of Tongji Hospital, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200802
Record Dates: First submitted 2020-08-02; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- spCART-269 (Experimental): spCART-269 administered by intravenous (IV) infusion
  Interventions: Biological: Targeting CD269 chimeric antigen receptor engineered T cells

INTERVENTIONS:
Biological: Targeting CD269 chimeric antigen receptor engineered T cells — Targeting CD269 chimeric antigen receptor engineered T cells, single infusion intravenously
  Other Names: spCART-269

SUMMARY:
The trial is a single arm, single-center, non-randomized phase I clinical trial which is designed to evaluate the safety and efficacy of spCART-269 in treatment of relapsed or refractory multiple myeloma patients.

DETAILED DESCRIPTION:
This study plans to enroll 10 patients to assess the safety and efficacy of spCART-269. Subjects who meet the eligibility criteria will receive a single dose of spCART-269 injection. The study will include the following sequential phases: Screening, Pre-treatment (Cell product preparation; Lymphodepleting Chemotherapy), Treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was diagnosed as active MM according to the diagnostic criteria of the International Myeloma Working Group (IMWG)
2. The patient meets any of the following:

   1. Have received at least 3 treatment options in the past and include alkylating agents, proteasome inhibitors and immunomodulators;
   2. If the patient has received a regimen containing proteasome inhibitor and immunomodulator for at least 2 courses, and the effect is not good (such as disease progression within 60 days of treatment)
3. Voluntary participation in clinical research and signing informed consent
4. Age 18-65, regardless of gender
5. Expected survival time is greater than 12 weeks
6. If the patient has received autologous hematopoietic stem cell transplantation in the past, a 90-day interval is required
7. Normal bone marrow hematopoietic function, blood routine: hemoglobin ≥ 100 g/L; absolute neutrophil ≥ 1.5×10^9/L; platelet count ≥ 100×10^9/L
8. Liver function: serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 (ULN) times the upper limit of normal value (if abnormal liver function is mainly caused by tumor infiltration, it can be ≤ 5 times the upper limit of normal value (ULN) )), bilirubin <2.0 mg/dL
9. Renal function: BUN is 9-20 mg/dL, serum creatinine ≤ 1.5 times the upper limit of normal (ULN), endogenous creatinine clearance rate ≥50 ml/min
10. Serum virus EBV, CMV, HBV, HCV, HIV and syphilis antibodies are negative
11. Heart function: good hemodynamic stability, left ventricular ejection fraction (LVEF) ≥ 45%
12. ECOG physical status score 0-2
13. Possess apheresis or sufficient venous access for venous blood, and no other contraindications for leukocyte separation
14. T cells can be successfully expanded in vitro
15. Women of childbearing age who provide negative reports of pregnancy tests with serum or urine before reinfusion
16. Adults with fertility requirements, regardless of sex, contraception within one year after treatment

Exclusion Criteria:

1. ECOG score ≥ 3 points
2. Female patients during pregnancy or lactation
3. Pathological examination revealed malignant tumor cells with T cell origin
4. Organ failure: Heart failure grade Ⅲ and Ⅳ; liver reaches Child-Turcotte liver function grade C; renal failure and uremia; respiratory failure; consciousness disorder
5. Patients with acute or chronic GVHD after allogeneic hematopoietic transplantation, or using hormones or immunosuppressants within 30 days
6. Patients with HIV infection or active hepatitis
7. There are other uncontrolled active infections
8. Those who may be allergic to cytokines
9. Those who have used any gene therapy products
10. Those who participated in other clinical studies 4 weeks before enrollment (except those who did not receive treatment in clinical studies)
11. Patients with systemic autoimmune diseases or immunodeficiency diseases
12. Definite neuropathy or psychosis, including authors of dementia or epilepsy
13. Those with lung or intestinal tumor infiltration
14. Patients that other researchers think are not suitable for enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | 12 weeks
  Incidence and severity of Treatment emergent adverse events

SECONDARY OUTCOMES:
Overall response rate (ORR) | 12 months
Duration of remission (DOR) | 12 months
Progression free survival (PFS) | 12 months
Overall survival (OS) | 12 weeks, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Aibin Liang, MD, Ph.D, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated and analysed during the current study are available from the corresponding author on reasonable request.